CLINICAL TRIAL: NCT03686917
Title: Validation of a CREATION Health Assessment Tool for Patients (CHAT-P) in a Diabetic Outpatient Population
Brief Title: Validation of a CREATION Health Assessment Tool for Patients in a Diabetic Outpatient Population
Acronym: CHAT-P
Status: Completed | Type: Observational
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 1304646
Record Dates: First submitted 2018-09-24; First posted 2018-09-27 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; type 2 diabetes; diabetes mellitus; type 2 diabetes mellitus; outpatient
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CHAT-P: Survey
  Interventions: Other: CHAT-P

INTERVENTIONS:
Other: CHAT-P — Survey

SUMMARY:
Participants will complete a survey before an educational session, during the "break" of an educational session, or after the session.

DETAILED DESCRIPTION:
Participants will be recruited from diabetes education sessions at selected locations and at FHMG physician practices. For the diabetes education setting, ta research team member will introduce this study to a group of patients before educational sessions, during "break" of the educational sessions, and after sessions. If the patient is interested, an envelope with the Invitation to Participant letter attached to it and the survey enclosed will be given to them. Also, a NOTE will be attached to the envelope with the instructions: "Please drop your completed survey in the drop-box at ___." The drop-box location will be identified within each setting and provided to the participants in the note or indicated verbally.

For patients at physician practices, an envelope with the Invitation to Participant letter attached to it and survey enclosed will be given by a staff member. Invitation to Participant letter contains all portions of the consent process. A NOTE will be attached to the envelope with the instructions: "Please drop your completed survey in the drop box at____." The drop-box location will be identified within each setting and provided to the participants in the note or indicated verbally. If patient does not meet the inclusion criteria, they will be asked to return the envelope to the staff member who provided it.

Patients will be provided with Invitation to Participate letter along with survey. The Invitation to Participate letter provides patients with study details including inclusion/exclusion criteria, duration of participation, procedures to ensure confidentiality, and an overview of voluntary participation conditions. Implied consent will be used. In addition to the Invitation to Participate letter, there is a statement at the top of the survey "return of completed surveys implies consent to participate in the study"

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and above
2. Diagnosis of type II diabetes
3. Able to speak and understand English
4. Able to provide informed consent

Exclusion Criteria:

1. Children under 18
2. Does not speak or understand English
3. Not of cognitive capacity to provide valid responses
4. Prisoners

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with type 2 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
CHAT-P Score | Survey administered one time at baseline during the single study visit.
  Total score of 28 item survey. Survey scored using a 5-point scale: Strongly disagree, Disagree, Neutral, Agree, Strongly Agree

SECONDARY OUTCOMES:
Demographics | Collected one time at baseline during the single study visit.
  Self reported demographics, including age, gender, and race
Adventist Wholeness Screening | Collected one time at baseline during the single study visit.
  4 item survey. Q1 is YES/NO. Q2-4 are Yes/No/Not Sure
Personal Wellbeing Index | Collected one time at baseline during the single study visit.
  9 items. Items are scored over an 11-point satisfaction scale with two response anchors of No Satisfaction at All / Completely Satisfied.
Multicultural Quality of Life Index | Collected one time at baseline during the single study visit.
  10 items, answers on a scale of 1-10, with one being "Poor" and 10 being "Excellent".

CONTACTS AND LOCATIONS:
Overall Officials: Hong Tao, PhD, Principal Investigator — AdventHealth
Locations (1):
- Center for Whole-Person Research, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Billioux, A., Verlander, K., Anthony, S., & Alley, D. (2017). Standardized screening for health-related social needs in clinical settings: The accountable health communities screening tool. Discussion Paper, National Academy of Medicine, Washington, DC. Retrieved from https://nam.edu/wp-content/uploads/2017/05/ Standardized-Screening-for-Health-Related-Social-Needsin-Clinical-Settings.pdf.
- [Background] Cummings, D., Reed, M., & Chobotar, T. (2015). Creation Health Discovery: Live Life to The Fullest (5th ed.). Maitland, FL: Florida Hospital Publishing.
- [Background] Polit, D. F. (2009) Data analysis & statistics for nursing research (2nd ed.). Upper Saddle River, NJ: Prentice Hall.
- [Background] Roozen HG, Wiersema H, Strietman M, Feij JA, Lewinsohn PM, Meyers RJ, Koks M, Vingerhoets JJ. Development and psychometric evaluation of the pleasant activities list. Am J Addict. 2008 Sep-Oct;17(5):422-35. doi: 10.1080/10550490802268678. PMID 18770086
- [Background] Stevens, J. (2002). Applied multivariate statistics for the social sciences (4th ed.). Mahwah, NJ: Lawrence Erlbaum Associates
- [Background] van Bokhorst-de van der Schueren MA, Guaitoli PR, Jansma EP, de Vet HC. Nutrition screening tools: does one size fit all? A systematic review of screening tools for the hospital setting. Clin Nutr. 2014 Feb;33(1):39-58. doi: 10.1016/j.clnu.2013.04.008. Epub 2013 Apr 19. PMID 23688831